CLINICAL TRIAL: NCT03222414
Title: Non-invasive Versus Invasive Blood Pressure Measurement in the Morbidly Obese Parturient (BMI >= 40 kg/m2) With Severe Preeclampsia: A Comparison of Direct Arterial Blood Pressure Measurements With Readings Obtained Using Either Large Cylindrical or Novel Conical Bariatric Upper Arm Blood Pressure Cuffs
Brief Title: Non-invasive Versus Invasive Blood Pressure Measurement in the Morbidly Obese Parturient With Severe Preeclampsia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Changes in standard of care have altered the feasibility of the study.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Laura Sorabella, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 150606
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Pre-Eclampsia; Morbid Obesity; Parturient; Blood Pressure
MeSH Terms: conditions — Pre-Eclampsia; Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A: Conical then Cylindrical (Experimental): BP recording with noninvasive conical Ultracheck Curve BP cuff and direct invasive arterial pressure monitoring; then with traditional cylindrical BP cuff and direct invasive arterial pressure monitoring
  Interventions: Device: Non-invasive BP recording with conical Ultracheck Curve BP cuff; Device: Non-invasive BP recording with traditional cylindrical BP cuff; Other: Direct invasive arterial pressure
- Arm B: Cylindrical then Conical (Active Comparator): BP recording with noninvasive traditional cylindrical BP cuff and direct invasive arterial pressure monitoring; then with conical Ultracheck Curve BP cuff and direct invasive arterial pressure monitoring
  Interventions: Device: Non-invasive BP recording with conical Ultracheck Curve BP cuff; Device: Non-invasive BP recording with traditional cylindrical BP cuff; Other: Direct invasive arterial pressure

INTERVENTIONS:
Device: Non-invasive BP recording with conical Ultracheck Curve BP cuff — Non-invasive SBP, DAP and MAP will be measured in both arms using conical Ultracheck Curve BP cuff
Device: Non-invasive BP recording with traditional cylindrical BP cuff — Non-invasive SBP, DAP and MAP will be measured in both arms using traditional cylindrical BP cuff
Other: Direct invasive arterial pressure — Direct invasive arterial pressure readings will be recorded simultaneously with non-invasive measurements

SUMMARY:
The study will compare agreement of invasive blood pressure measurements with non-invasive blood pressure measurements measured with a conical blood pressure and large standard upper arm rectangular cuff in morbidly obese severely hypertensive (systolic blood pressure > 160 mmHg) parturients.

DETAILED DESCRIPTION:
A morbidly obese [Body Mass Index (BMI) ≥ 40 kg/m2] pregnant woman is at singular risk for all the complications of pregnancy, most notably preeclampsia (PE). Furthermore a woman who is already chronically hypertensive is likely to develop superimposed PE . Uncontrolled systolic hypertension in pregnancy prompts placental abruption, hemorrhagic stroke, and systolic or diastolic heart failure. Accurate blood pressure measurement is therefore a prerequisite to controlling dangerously high systolic blood pressure (SBP) to enable labor and delivery to be conducted safely in association with PE. Precise SBP measurement is also a precondition for clinically testing hypotheses concerning the existence of druggable targets that will allow prolongation of pregnancy in the face of severe PE and /or intra-uterine growth restriction (IUGR) remote from term.

Oscillometric noninvasive blood pressure (NIBP) measurement is the customary standard blood pressure monitoring method most often used in the labor suite and obstetric operating room today. For this purpose a rectangular, cylindrical blood pressure (BP) cuff placed on the upper arm is connected to an oscillometric blood pressure device. Yet inaccuracies related to the fact that oscillometric NIBP devices under-read high SBP relative to IBP measurements have been recognized as a potential source of maternal morbidity for years.

The study will compare IBP readings obtained from morbidly obese, severely hypertensive (SBP > 160 mm Hg) parturients with NIBP consecutively measured with new innovative conical Ultracheck Curve BP cuffs and large standard upper arm rectangular cylindrical BP cuffs.

ELIGIBILITY:
Inclusion Criteria:

* Written, signed and dated informed consent
* ≥ 18 years of age
* BMI >40 kg/m2
* Has a clinically indicated radial artery line already in situ or who agree to placement of an arterial line
* Systolic blood pressure >160 mm Hg
* Gestational age greater than or equal to 24 weeks
* Parturients admitted for induction of labor

Exclusion Criteria:

* Parturients admitted in labor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-01-18 (Actual); Study Completion 2016-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sorabella, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ashworth DC, Maule SP, Stewart F, Nathan HL, Shennan AH, Chappell LC. Setting and techniques for monitoring blood pressure during pregnancy. Cochrane Database Syst Rev. 2020 Jul 23;8(8):CD012739. doi: 10.1002/14651858.CD012739.pub2. PMID 32748394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were randomized, but data was not analyzable on 2 participants. Randomization assignment was not recorded on these 2 participants.
Period: Overall Study
Arm/Group | Arm A: Conical Then Cylindrical | Arm B: Cylindrical Then Conical
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 3 participants were randomized, but data was collected incorrectly on 2 participants, so data was unusable on those 2 participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Conical Then Cylindrical | Arm B: Cylindrical Then Conical | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Noninvasive Systolic Blood Pressure Readings to Invasive Blood Pressure Measurement
Description: Absolute difference between the mean of 2 non-invasive systolic blood pressure readings and mean of 2 invasive systolic blood pressure readings
Time Frame: Single time point measurement (1 day)
Measure: Number; unit: mm Hg
Groups:
- Conical: BP recording with noninvasive conical Ultracheck Curve BP cuff and direct invasive arterial pressure monitoring;
  Non-invasive BP recording with conical Ultracheck Curve BP cuff: Non-invasive SBP, DAP and MAP will be measured in both arms using conical Ultracheck Curve BP cuff
  Direct invasive arterial pressure: Direct invasive arterial pressure readings will be recorded simultaneously with non-invasive measurements
- Cylindrical: Non-invasive BP recording with traditional cylindrical BP cuff: Non-invasive SBP, DAP and MAP will be measured in both arms using traditional cylindrical BP cuff
  Direct invasive arterial pressure: Direct invasive arterial pressure readings will be recorded simultaneously with non-invasive measurements
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | -28 | -6.5

2. Secondary Outcome: Comparison of Mean Arterial Pressure (MAP) Measured Withnon-invasive Cuffs to MAP Measured by Invasive Blood Pressure Monitoring
Description: Absolute difference in the mean of 2 non-invasive MAP readings and mean of 2 invasive MAP readings
Time Frame: Single time point measurement (1 day)
Measure: Number; unit: mm Hg
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | -25 | -13.5

3. Secondary Outcome: Comparison of Noninvasive Diastolic Blood Pressure Readings to Invasive Blood Pressure Measurement
Description: Absolute difference between the mean of 2 non-invasive diastolic blood pressure readings and mean of 2 invasive diastolic blood pressure readings
Time Frame: Single time point measurement (1 day)
Measure: Number; unit: mm Hg
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | -9.5 | 0.5

4. Secondary Outcome: Mean of 2 Systolic Blood Pressure Readings Taken With Cylindrical and Conical BP Cuffs
Description: mean of 2 systolic blood pressure readings taken with cylindrical and conical BP cuffs
Time Frame: Single time point measurement (1 day)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | 132.5 (2.12) | 154 (1.41)

5. Secondary Outcome: Mean of 2 MAP Readings Taken With Cylindrical and Conical BP Cuffs
Description: Mean of 2 MAP readings taken with cylindrical and conical BP cuffs
Time Frame: Single time point measurement (1 day)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | 87.5 (2.12) | 101.5 (0.71)

6. Secondary Outcome: Mean of 2 Diastolic Blood Pressure Non-invasive BP Measurements Taken With Cylindrical and Conical BP Cuffs
Description: Mean of 2 diastolic blood pressure non-invasive BP measurements taken with cylindrical and conical BP cuffs
Time Frame: Single time point measurement (1 day)
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Conical | Cylindrical
Number analyzed (Participants) | 1 | 1
mm Hg | 73.5 (3.54) | 85 (2.83)

ADVERSE EVENTS:
Time Frame: 1 hour
Description: there were 0 in that arm
Arm/Group | Arm A: Conical Then Cylindrical | Arm B: Cylindrical Then Conical
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/14/NCT03222414/Prot_SAP_000.pdf